CLINICAL TRIAL: NCT05896826
Title: Ultra-sensitive Magnetocardiography in the Accurate Identification of Myocardial Infarction
Brief Title: Magnetocardiography in the Accurate Identification of Myocardial Infarction
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Chongqing Emergency Medical Center (Other); Weifang People's Hospital (Other); Linyi People's Hospital (Other); Weihai Central Hospital (Other); Jining First People's Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Qianfoshan Hospital (Other); Heze Municipal Hospital (Other); First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Other Study IDs: QLEmer-MCG
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Chest Pain; Acute Coronary Syndrome; Myocardial Infarction
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy volunteers
  Interventions: Device: Magnetometer
- chest pain patients who will receive ECG, biomarkers, or non-invasive imaging examination
  Interventions: Device: Magnetometer

INTERVENTIONS:
Device: Magnetometer — inspection equipment for magnetocardiography

SUMMARY:
Magnetocardiography (MCG) is a promising noninvasive and accurate method for detecting myocardial infarction. Although progress has been made in this area, there is a lack of studies using up-to-date examination instruments for the calibration of MCG analysis. This is a prospective single-center study aiming to build accurate analytical models of MCG to detect myocardial infarction. Myocardial infarction are diagnosed by electrocardiogram, biomarkers (high-sensitivity cardiac troponin, etc), or non-invasive imaging (cardiac magnetic resonance or single-photon-emission tomography). Myocardial infarction is also quantified by cardiac magnetic resonance or single-photon-emission tomography. Healthy volunteers and chest pain patients who will receive electrocardiogram, biomarkers (high-sensitivity cardiac troponin, etc), or non-invasive imaging (cardiac magnetic resonance or single-photon-emission tomography) examination will be enrolled in this study.

ELIGIBILITY:
For healthy volunteers:

Inclusion Criteria:

1. Age 18-79 years old;
2. No history of cardiovascular disease (coronary heart disease, structural heart disease, arrhythmia, heart failure, stroke, pulmonary embolism, aortic dissection, etc.), no cardiovascular risk factors (hypertension, diabetes, hyperlipidemia). For people over 65 years old, those with hypertension or hyperlipidemia, but with well-controlled blood pressure and lipid levels, taking no more than 2 drugs, and echocardiography showing no left ventricular hypertrophy, can be included;
3. The electrocardiogram is normal, and the cardiac ultrasound is basically normal in the past 1 year (mild valvular regurgitation can be included).
4. Sign the informed consent.

Exclusion Criteria:

1. Those who with acute or chronic respiratory diseases;
2. Those who with obvious abnormality of liver or kidney function;
3. Those who with endocrine diseases such as abnormal thyroid function;
4. Those who with anemia or other blood diseases;
5. Those who with connective tissue diseases (lupus erythematosus, rheumatoid arthritis, dermatomyositis, polyarteritis nodosa, etc.);
6. Those who are obese (BMI>30kg/cm2) or underweight (BMI<18kg/cm2);
7. Those who with malignant tumors;
8. Those who with infectious diseases or infectious diseases;
9. Those who with trauma or physical disability;
10. Those who with psychological or mental illness such as depression;
11. Those who are professional athletes, pregnant or breastfeeding women, alcoholics;
12. Those who are unable to perform magnetocardiography examination due to claustrophobia, etc., or those who fail to receive magnetocardiography examination;
13. Due to various reasons such as allergy to contrast agents, metal implants in vivo that are prohibited from performing 1.5T MRI (such as prostheses or steel plates implanted in orthopaedics, uterine contraceptive device) and other reasons, those who cannot or fail to cooperate with the corresponding research requirements.

For chest pain patients who will receive ECG, biomarkers, or non-invasive imaging examination:

Inclusion Criteria:

1. Age 18-79 years old;
2. Those with chest pain symptoms, diagnosed or highly suspected by the attending doctor or above as stable angina pectoris (SA), unstable angina pectoris (UA), non-ST segment elevation myocardial infarction (NSTEMI), ST segment elevation myocardial infarction (STEMI), and plan to receive electrocardiogram, biomarkers (high-sensitivity cardiac troponin, etc), or non-invasive imaging (cardiac magnetic resonance or single-photon-emission tomography);
3. Sign the informed consent.

Exclusion Criteria:

1. Patients with known structural heart disease such as cardiomyopathy and valvular disease;
2. Patients with arrhythmias such as atrial fibrillation, supraventricular tachycardia, and atrioventricular block that have not returned to normal;
3. History of other cardiovascular diseases such as pulmonary embolism and aortic dissection;
4. Patients with connective tissue diseases (lupus erythematosus, rheumatoid arthritis, dermatomyositis, polyarteritis nodosa, etc.) combined with cardiac complications;
5. Obvious abnormal thyroid function, severe anemia or other blood diseases and other diseases that obviously affect the circulating blood supply;
6. Obese (BMI>30kg/cm2) or underweight (BMI<18kg/cm2);
7. Patients with malignant tumors;
8. Professional athletes, pregnant or breastfeeding women, alcoholics;
9. Acute diseases or critical illnesses in other systems, such as acute or severe respiratory diseases, abnormal liver function or renal function, etc.;
10. Patients with infectious diseases or infectious diseases;
11. Those who are unable or fail to perform magnetocardiography due to claustrophobia, physical impairment, etc.;
12. Unable to or fail to cooperate with the corresponding research requirements.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy individuals and chest pain patients who will receive ECG, biomarkers, or non-invasive imaging examination
Sampling Method: Non-Probability Sample
Enrollment: 3841 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of MCG to detect myocardial infarction | 6 hours
  To establish an algorithm model of MCG in detecting myocardial infarction and to assess the sensitivity and specificity of the above model in detecting myocardial infarction. Myocardial infarction are diagnosed by electrocardiogram, biomarkers (high-sensitivity cardiac troponin, etc), or non-invasive imaging (cardiac magnetic resonance or single-photon-emission tomography).

SECONDARY OUTCOMES:
Accuracy of MCG to detect the localization of myocardial infarct | 6 hours
  To build up an algorithm model of MCG in detecting the localization of myocardial infarct. The sensitivity and specificity of the model in detecting infarct location were evaluated.
Accuracy of MCG in identifying myocardial infarct sizes | 6 hours
  To establish an algorithm model of MCG in detecting identifying myocardial infarct sizes and to assess the sensitivity and specificity of the above model in identifying myocardial infarct sizes. Myocardial infarction sizes is quantified by cardiac magnetic resonance or single-photon-emission tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguo Chen, Dr, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China